CLINICAL TRIAL: NCT01531959
Title: Midodrine for the Treatment of Refractory Hypotension in Patients Otherwise Ready for Discharge From the ICU
Brief Title: Midodrine for the Treatment of Refractory Hypotension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sir Charles Gairdner Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, MD PhD, Vice Chair of Faculty Affairs of the Department of Anesthesia Critical Care and Pain Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011P002049; 2015-098 (Other: Sir Charles Gairdner Hospital HREC); 2018P000162 (Other: Beth Israel Deaconess Medical Center)
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Hypotension; Critical Illness
Keywords: Midodrine; Hypotension; Intensive care unit; IV vasopressors; ICU discharge
MeSH Terms: conditions — Hypotension; Critical Illness | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midodrine (Active Comparator)
  Interventions: Drug: Midodrine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine — Patients will be randomized to blinded to 20 mg of midodrine
  Arms: Midodrine
Drug: Placebo — Patients will be randomized to blinded placebo control
  Arms: Placebo

SUMMARY:
We hypothesize that midodrine treatment of refractory hypotension in patients otherwise ready for discharge from the ICU shortens duration of receiving IV vasopressors and SICU length of stay without increasing MGH length of stay or putting the patient at risk of being readmitted to an ICU.

DETAILED DESCRIPTION:
Persistent hypotension in critically ill patients remains a major barrier to discharging patients from the intensive care unit (ICU). In our hospital, in patients with adequate tissue perfusion, midodrine has been observed to treat hypotension in order to wean continuous intravenous (IV) vasopressors and therefore promote ICU discharge. There are several possible etiologies of hypotension in the ICU. The most frequently seen causes include septic shock, hypovolemia, adrenal insufficiency, and idiosyncratic reactions from medications. For patients whose reversible causes of hypotension have been addressed but still require vasopressors, midodrine may prove to be a useful adjunctive medication to successfully increase blood pressure. No previous studies have examined the use of midodrine for the treatment of hypotension in an ICU setting. Therefore, we are investigating a new indication for midodrine as the treatment of hypotension in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Admitted to the SICU
* Requiring IV vasopressors at a rate of less than 100 mcg/min of phenylephrine, or 8 mcg/min of norepinephrine, or 60 mcg/min of metaraminol; and unable to wean for more than 24 hours while still maintaining desired blood pressure goal

Exclusion Criteria:

* Inadequate tissue oxygenation
* Liver failure
* Renal failure
* Hypovolemic shock or hypotension due to adrenal insufficiency
* Pregnancy
* Severe organic heart disease
* Urinary retention
* Pheochromocytoma
* Thyrotoxicosis
* Midodrine as pre-admission medication
* Any known allergies to midodrine
* Enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-04; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia

REFERENCES:
- [Derived] Anstey MH, Wibrow B, Thevathasan T, Roberts B, Chhangani K, Ng PY, Levine A, DiBiasio A, Sarge T, Eikermann M. Midodrine as adjunctive support for treatment of refractory hypotension in the intensive care unit: a multicenter, randomized, placebo controlled trial (the MIDAS trial). BMC Anesthesiol. 2017 Mar 21;17(1):47. doi: 10.1186/s12871-017-0339-x. PMID 28327122

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 139 participants provided informed consent and were enrolled. 3 participants subsequently did no loner meet eligibility criteria and were therefore not randomized, resulting in a total number of started/randomized participants of 136.
Period: Overall Study
Arm/Group | Midodrine | Placebo
Started | 68 | 68
Completed | 66 | 66
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midodrine | Placebo | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (12.6) | 66.7 (14.7) | 68.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 36 | 32 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 62 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
APACHE II Score [Mean (Standard Deviation); unit: units on a scale] — The Acute Physiology and Chronic Health Evaluation (APACHE II) score is an mortality prediction score used in critically ill patients. I ranges from 0 (minimum) to 71 (maximum), with lower score values representing better outcomes.
  units on a scale | 14.7 (5.2) | 14.8 (5.9) | 14.7 (5.5)
SOFA Score on admission day [Median (Inter-Quartile Range); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) score is a score that allows for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic). I ranges from 0 (minimum) to 24 (maximum), with lower score values representing better outcomes.
  units on a scale | 4 [3 to 5] | 5 [3 to 7] | 4 [3 to 6]
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (8.8) | 29.8 (8.8) | 28.8 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Time Until Discontinuation of IV Vasopressors
Description: Measured hours from initiation of midodrine until discontinuation of IV vasopressors
Time Frame: From initiation of the study drug until discontinuation of IV vasopressors, assessed up to 400 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 66 | 66
hours | 23.5 [10.0 to 54.0] | 22.5 [10.4 to 40.0]

2. Secondary Outcome: ICU Length of Stay
Description: Measured number of days from initiation of midodrine until discharge ready from the ICU
Time Frame: From initiation of midodrine until ICU discharge, assessed up to 45 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 66 | 66
days | 6.0 [5.0 to 8.0] | 6.0 [4.0 to 8.0]

3. Secondary Outcome: Hospital Length of Stay
Description: Measured number of days from initiation of midodrine until discharged from hospital
Time Frame: From initiation of midodrine until hospital discharge, assessed up to 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 66 | 66
days | 11.0 [9.0 to 21.0] | 14.0 [9.0 to 22.0]

4. Secondary Outcome: Rates of ICU Readmission
Description: Number of patients initiated on midodrine that are readmitted back to ICU after being discharged to floor
Time Frame: Up to 2 months after ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 66 | 66
Participants | 1 | 3

5. Secondary Outcome: Rates of Hypertension, Bradycardia, and Hemodynamically Significant Tacharrythmias
Description: Measured rates of hypertension (increase in systolic blood pressure to values higher than those set by the primary team or greater than 160 mmg), bradycardia (decrease in heart rate to values lower than those set by the primary team or less than 40 BPM), hemodynamically significant tachyarrythmias (greater than 20 mmhg decrease in systolic blood pressure).
Time Frame: From initiation of the study drug until discontinuation of the study drug, an average of 59 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 66 | 66
Participants | 12 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected daily from medical records for the period of study drug administration, an average of 59 hours.
Arm/Group | Midodrine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/66 | 1/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/66
Other Adverse Events (participants affected / at risk) | 20/66 | 17/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midodrine (N=66) | Placebo (N=66)
Death (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midodrine (N=66) | Placebo (N=66)
Hypertension (Cardiac disorders) | 7 (7) | 3 (3)
Bradycardia (Cardiac disorders) | 5 (5) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Lab parameter change (Investigations) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough/dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Myocardial infarction/ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Peripheral edema (General disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular ectopic beats (Cardiac disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Subdural hemtoma (Nervous system disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT01531959/Prot_SAP_000.pdf